CLINICAL TRIAL: NCT00226148
Title: Immediate Implant Placement in the Molar Regions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Thomas Urban, Dental School, Aarhus University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/0091; 22-04-0281
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Periodontitis; Dental Caries; Periapical Periodontitis
Keywords: Implant; Immediate placement; Molar tooth
MeSH Terms: conditions — Periodontitis; Dental Caries; Periapical Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Use of a membrane to cover bonedefects around implant
Device: Use of bonechips to fill up defects around implant
Procedure: Use of membrane and bonechips to manage defects

SUMMARY:
The purpose of this study is to look at the bonehealing when a molar has been extracted and immediately replaced by an implant leaving some defects around the implant.

The defects are being treated in three different with the hypothesis that the three ways of treatment result in equal bonehealing.

DETAILED DESCRIPTION:
This study is a randomized clinically controlled study with three group of each thirty patients, where the bonehealing after immediate implantplacement in molarregions is being investigated.

Totally 90 patients are going to get a molar tooth extracted and immediately replaced with an implant (Brånemark System, Wide Platform). The molar tooth should be in such a condition that is has to be extracted.

Extracting a molar leaves a defect which cannot completely be filled out by an implant. The 90 patients are therefore randomised into 3 groups according to how the perimarginal bonedefects around the placed implants are being treated: 1. Bonechips 2. Membrane 3. Bonechips+Membrane. The bonehealing of the defects around the implants are then compared the groups in between. The amount of newly formed bone is being estimated too by digital radiography and subtractionradiography. Furthermore the prognosis for immediate placed implants in molar regions in relation to the method of defectreconstruction one year after crown delivery is also being investigated. All the investigations are conducted with the Ho-hypothesis that there is no difference in the bonehealing the three groups in between.

ELIGIBILITY:
Inclusion Criteria:

* A molar tooth which has to be extracted
* Healthy persons with only mild systemic disease with no functional limitation

Exclusion Criteria:

* Pregnant
* Any disease that is influencing the turnover of bone or oral mucosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Digitial radiography of the implants at placement, 3 month, 6 month, at abutmentoperation, at crownplacement, 3 month after crownplacement and 6 month after crownplacement. | see above

CONTACTS AND LOCATIONS:
Overall Officials: Ann Wenzel, Prof.Dr.Odont, Ph.d.,DDS, Study Chair — The Royal Dental College of Aarhus
Locations (1):
- The Royal Dental College of Aarhus, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Urban T, Kostopoulos L, Wenzel A. Immediate implant placement in molar regions: a 12-month prospective, randomized follow-up study. Clin Oral Implants Res. 2012 Dec;23(12):1389-97. doi: 10.1111/j.1600-0501.2011.02319.x. Epub 2011 Nov 25. PMID 22117841